CLINICAL TRIAL: NCT03456206
Title: Intake of Dietary Fibre, Red and Processed Meat and Risk of Late-Onset Chronic Inflammatory Diseases: A Prospective Danish Study on the "Diet, Cancer and Health" Cohort
Brief Title: Chronic Inflammatory Disease, Lifestyle and Risk of Disease
Acronym: PROCID-DCH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Hospital of Southern Jutland (Other); Odense Patient Data Explorative Network (Other); University of Aarhus (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Vibeke Andersen, Professor, University of Southern Denmark
Other Study IDs: PROCID-DCH
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Autoimmune Diseases; Inflammatory Bowel Diseases; Crohn Disease (CD); Ulcerative Colitis (UC); Arthritis, Rheumatoid (RA); Spondylarthropathies; Arthritis, Psoriatic (PsA); Psoriasis (PsO); Multiple Sclerosis (MS)
Keywords: Life Style; Diet; Food; CID; Disease risk
MeSH Terms: conditions — Autoimmune Diseases; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Spondylarthropathies; Arthritis, Psoriatic; Psoriasis; Multiple Sclerosis | interventions — Dietary Fiber

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "Diet, Cancer and Health" cohort: Participants from the "Diet, Cancer and Health" (DCH) cohort with no CID diagnosis at entry to the DCH study. The number of persons developing a CID (defined as at least one of the mentioned CIDs) during follow up (1993/1997 - 2018) and the number of persons not developing a CID will be investigated.
  Based on the participants reporting of dietary habits in the Food Frequency Questionnaire (FFQ) from the DCH study, the exposure "intake of red and processed meat and fibres" will be investigated in both CID cases and non-cases.
  Other exposure variables are "Lifestyle factors independently or combined" and are also obtained from the data in the DCH cohort.
  Interventions: Other: Intake of red and processed meat and fibres; Other: Lifestyle factors independently or combined

INTERVENTIONS:
Other: Intake of red and processed meat and fibres — The intention is to analyse exposure groups in tertiles: 1) Upper tertile (33.3% of the total sample) based on the ratio: meat/fibre intake is associated with higher risk of CID. 2) Low intake of fibre (defined as below the lower tertile [33.3% of the total sample]) and high intake of red and processed meat (defined as those above the upper tertile [33.3% of the total sample]) are independently associated with higher risk of CID, and their synergy (interaction between the factors meat and fibres) gives the highest risk outcome.
Other: Lifestyle factors independently or combined — Lifestyles factors are defined as: red and processed meat, vegetables, dietary fibre, cereals, gluten, legumes, red wine, dairy products, physical activity, smoking, total protein/fat, protein/fat from red and processed meat, glycemic index.

SUMMARY:
Chronic inflammatory diseases (CID) - including inflammatory bowel diseases (Crohn's disease and ulcerative colitis), rheumatic conditions (rheumatoid arthritis, axial spondyloarthritis, psoriatic arthritis), inflammatory skin diseases (psoriasis) and multiple sclerosis are diseases of the immune system that have some shared genetic and environmental predisposing factors, but still little is known on the effects of lifestyle as a prognostic factor on disease risk. This observational study will contribute to preexisting research on lifestyle factors by identifying diet factors associated with risk of developing CID, using prospective register data.

The study will use data from all of the 57,053 participants in the Danish cohort "Diet, Health and Cancer (DHC)" together with registry data. Blood samples, anthropometric measures and questionnaire data on diet and lifestyle were collected at the DHC study entry. The National Patient Registry (NPR) will be used to obtain to identify patients with CID during follow-up. Follow-up information on death and immigration will be collected in March 2018 from the Danish Civil Registration Register.

The outcome CID is defined as at least one of the following CIDs: Crohn's disease, ulcerative colitis, psoriasis/psoriatic arthritis, rheumatoid arthritis/ankylosing arthritis, or multiple sclerosis, during the follow-up period from 1993 to March 2018.

The primary hypothesis is that "the risk of CID will be significantly higher among those with a low fibre/high red and processed meat intake compared to those with a high fibre/low red and processed meat intake." Based on previous research on a shared etiology in CIDs a second hypothesis is that "the postulated causality between low fibre/high red and processed meat intake and risk of developing CID is applicable for each of the CID-diagnoses."

The core study is an open register-based cohort study. The study does not need approval from the local Ethics committee or Institutional Review Board by Danish law. The study was approved by the Danish Data Protection Agency (2012-58-0018) Study findings will be disseminated through peer-reviewed journals, patient associations and presentations at international conferences.

DETAILED DESCRIPTION:
Material and methods:

The study design is a cohort study with prospective register data follow up. The Danish cohort "Diet, Health and Cancer" (DHC) will be used. The DHC Study is an ongoing Danish cohort study designed to investigate the relation between diet, lifestyle and disease risk. The cohort consists of 57,053 persons, recruited between December 1993 and May 1997. All the subjects (50 to 64 years of age) gave detailed information on diet (food frequency questionnaire) and other lifestyle data together with biological samples. Blood samples, anthropometric measures and questionnaire data on diet and lifestyle were collected at study entry. Data from the DHC cohort will be combined with Danish national registers (the National Patient Registry (NPR), the Danish Civil Registration Register, and The Danish National Prescription Registry).

Outcome measures and follow-up: The National Patient Registry (NPR) will be used to obtain to identify patients with CID during follow-up. The NPR contains data on all patients admitted to Danish hospitals since 1977. The register covers both inpatient and outpatient records and indicates the main medical reason for diagnostic procedures or treatment (since 1994 according to the tenth version of the International Classification of Diseases (ICD-10)). For this study there will be extracted data from NPR from 1993 to March 2018. The outcome CID is defined as at least one of the following diseases in the NPR; inflammatory bowel disease (IBD) (ICD10 codes: K50-K51), psoriasis/psoriatic arthritis (ICD10 codes: M073, M090, L40), rheumatoid arthritis/ankylosing arthritis (ICD10 codes: M059. M060, M069, M089, M459, M46), or multiple sclerosis (ICD10 codes: G35, G35.9), during the follow-up period. The Danish National Prescription Registry will be used to identify the most severe cases of the following diseases listed above, as it is expected that the patients have medication in relation to the diseases. Follow-up information on death and immigration will be collected in March 2018 from the Danish Civil Registration Register.

Exposure and possible confounders: Information on exposure is defined as high fibre intake and high red and processed meat intake and were collected at enrolment of the DHC cohort using questionnaires and interviews. In short, the food-frequency questionnaire, diet consumption was assessed in 12 categories of predefined responses, ranking from "never" to "eight times or more per day". The daily intake was then calculated by the software program FoodCalc. FoodCalc is a simple program to calculate intake of nutrients when given a list with amounts of different foods consumed and another list with contents of nutrients for the different foods. Both intake of dietary fibre and red meat and processed meat were measured as continues variable in g/day. Information on possible confounders will also be obtained from the questionnaire data at enrolment in relation to sex, age, BMI, smoking and other lifestyle factors and information on co-morbidity will be obtained from NPR.

Statistical analyses: The intention is to use data obtained from this prospective cohort study to explore the ability to predict risk of CID (Y=primary endpoint) and to explore whether diets low in fibre AND high in red and processed meat (X=assessed at baseline) are an informative prognostic factor on disease risk. Descriptive analyses for categorical variables will be presented as frequencies, and differences between CID cases and non-cases will be evaluated by Chi-square test. Continuous variables will be tabulated as medians (with quartiles, Q1 and Q3) and nonparametric tests on the equality of medians will be used to test for differences between groups. P-values below 0.05 will be considered statistically significant. Negative binomial regression will be applied to calculate incidence rates per 1000 patient years and incidence rate ratios (IRR) between exposures. To investigate the risk of and time to CID-diagnosis the Fine-Gray competing risk regression model will be applied, and thus competing risk of death will be taken into account while handling emigration as censoring, and reporting cumulative incidences and sub-hazard ratios (SHR) and the corresponding p-values for CID associated with specified food substitutions. Regressions will be carried out as both crude regression, only including the exposure, and adjusted for age, sex, lifestyle factors and selected comorbidities. Analyses will be conducted using Stata.

To test if the hypothesized causality between diet factors and development of CID is applicable for all of the CIDs there will be conducted subanalyses on each of the CID-diagnoses. Sensitivity analyses will be conducted on data from the Danish National Prescription Registry to evaluate the validity of the CID diagnoses, as it is expected that they get treatment in relation to the diseases. Data on medication and treatment of each diagnosis will be analysed separately.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the DHC cohort

Exclusion Criteria:

* Participant with a CID diagnosis at entry

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All 57,053 participants from the DHC cohort
Sampling Method: Probability Sample
Enrollment: 57053 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
CID diagnosis | 24-28 years
  * Crohn's disease (yes/no)
  * Ulcerative colitis (yes/no)
  * Rheumatoid arthritis (yes/no)
  * Axial spondyloarthritis (yes/no)
  * Psoriatic arthritis (yes/no)
  * Psoriasis (yes/no)
  * Multiple sclerosis (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Andersen, Prof, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen NF, Rubin KH, Stougaard M, Tjonneland A, Stenager E, Lund Hetland M, Glintborg B, Bygum A, Andersen V. Impact of red meat, processed meat and fibre intake on risk of late-onset chronic inflammatory diseases: prospective cohort study on lifestyle factors using the Danish 'Diet, Cancer and Health' cohort (PROCID-DCH): protocol. BMJ Open. 2019 Mar 30;9(3):e024555. doi: 10.1136/bmjopen-2018-024555. PMID 30928934
- See also: Intake of dietary fibre, red and processed meat and risk of late-onset Chronic Inflammatory Diseases: A prospective Danish study on the "diet, cancer and health" cohort — https://pubmed.ncbi.nlm.nih.gov/33029091/